CLINICAL TRIAL: NCT05420779
Title: A Randomized, Parallel, Open-label, Positive Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of TSL-1502 Capsules in HER2-negative Locally Advanced or Metastatic Breast Cancer Patients With Germline BRCA Mutations
Brief Title: A Study to Evaluate the Efficacy and Safety of TSL-1502 Capsules in Breast Cancer Patients With Germline BRCA Mutations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Tasly Diyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Tasly Pharmaceutical Group Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSL-CM-TSL1502-Ⅱ
Record Dates: First submitted 2022-05-22; First posted 2022-06-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Metastatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TSL-1502 low dose group (Experimental): TSL-1502 capsules 350 mg,qd,po
  Interventions: Drug: TSL-1502 capsules(low dose)
- TSL-1502 high dose group (Experimental): TSL-1502 capsules 500 mg,qd,po
  Interventions: Drug: TSL-1502 capsules(high dose)
- Positive control group (Active Comparator): Investigator selects chemotherapy regimens according to the subjects' conditions.
  Interventions: Drug: Investigator's choice of chemotherapy

INTERVENTIONS:
Drug: TSL-1502 capsules(low dose) — 350 mg each time, orally administered QD, every 3 weeks as a treatment cycle.
  Arms: TSL-1502 low dose group
Drug: TSL-1502 capsules(high dose) — 500 mg each time, orally administered QD, every 3 weeks as a treatment cycle.
  Arms: TSL-1502 high dose group
Drug: Investigator's choice of chemotherapy — Capecitabine tablets, 1250 mg/m2 each time, BID oral administration; Vinorelbine tartrate injection, 25 ~ 30 mg/m2 each time, intravenous drip (15 ~ 20 min); Eribulin mesylate injection, 1.4 mg/m2 each time, intravenous injection (2 ~ 5 min)
  Arms: Positive control group

SUMMARY:
This research study is evaluating the efficacy and safety of TSL-1502 capsules in patients with breast cancer, will be included HER2-negative locally advanced or metastatic breast cancer patients with germline BRCA mutations.

DETAILED DESCRIPTION:
Background:

Breast cancer is a collective term for a variety of malignant breast tumors.According to the World Cancer Report newly released by the World Health Organization in February 2020, breast cancer ranks first in the causes of death among women due to cancer worldwide, with about 2.1 million new cases and 627,000 deaths in 2018. At present, the main treatments for breast cancer are surgery, chemotherapy, and endocrine therapy, but the therapeutic effect is limited. The 5-year survival rate for patients with advanced breast cancer is only 20%, and the overall survival (OS) is 2 ~ 3 years.

Research basis:

Tumor cells can activate their own DNA repair machinery to repair DNA damage caused by drugs and thus become resistant to radiotherapy and chemotherapy, while there is overexpression of DNA repair enzymes in a variety of tumor cells. Therefore, reducing the expression of DNA repair enzymes or inhibiting their activity may exert latent anti-tumor effects.

Specific aims:

To evaluate the objective response rate at least 4 weeks later,disease control rate,duration of response,progression-free survival and objective response rate and overall survival in patients withHER2-negative locally advanced or metastatic breast cancer patients with germline BRCA mutations. Also we plan to estimate safety endpoints and PK endpoints in this subject population.

Treatment plan:

Patients will be randomized in three arms. In arm A , patients will be treated with low dose TSL-1502 capsules, 350 mg each time, orally administered QD, every 3 weeks as a treatment cycle. In arm B , patients will be treated with the same interference with high dose,500 mg each time, orally administered QD, every 3 weeks as a treatment cycle. In arm B , patients will be treated with investigator's choice of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1) Agree to follow the clinical trial protocol, volunteer, and sign the informed consent form (ICF).

  2) Women aged ≥ 18 years and ≤ 75 years at the date of signing the ICF. 3) HER2-locally advanced breast cancer diagnosed by histopathology and/or cytology (Unable to receive radical therapy) or metastatic breast cancer, and previous chemotherapeutic line of cytotoxicity for locally advanced or metastatic breast cancer was ≤ 3.

  4) Prior platinum therapy is allowed, but the best response to platinum therapy is required to be CR, PR, or persistent ≥ 12 weeks SD. If given as neoadjuvant/adjuvant therapy, the time from the last dose of platinum to relapse is ≥ 6 months.

  5) Hormone receptor-positive patients need to have received at least first-line of endocrine therapy for locally advanced or metastatic breast cancer but failed, or unsuitable for endocrine therapy in the judgment of the investigator.

  6) In neoadjuvant, adjuvant and/or metastatic stages, the patients who have received antitumor therapy with Taxane ± Anthracycline.

  7) Failure of front-line therapy (disease progression or toxicity intolerance), and the investigator judged that it was suitable to receive the systemic monotherapy (including capecitabine tablets, vinorelbine tartrate injection, eribulin mesylate injection).

  8) Tested or reviewed by a third-party central laboratory to determine whether there is harmful or suspected harmful gBBRCAm in the blood.

  9) At least one measurable (non-lymph node longest diameter ≥ 10 mm, lymph nodes with a minimum diameter of ≥ 15 mm, according to RECIST version 1.1 criteria) of target lesions. Note: Previously irradiated lesions cannot be used as targets lesions unless there is significant progression of the lesion.

  10) The physical condition score is 0-1 according to the scale of The Eastern Cooperative Oncology Group (ECOG).

  11) Expected survival ≥ 12 weeks. 12) Meet the following criteria (The use of any blood components and cell growth factors is not permitted within 2 weeks prior to initial administration): Bone marrow function: absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1500/mm3); platelets ≥ 100 × 109/L (1 × 105/mm3); Hemoglobin ≥ 90 g/L; Liver function: serum bilirubin ≤ 1.5 × upper limit of normal (ULN), but except for Gilbert's syndrome patients (persistent or recurrent hyperbilirubinemia, unbound bilirubin elevation is present in the absence of evidence of hemolysis or liver pathology); patients without liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; ALT and AST ≤ 5×ULN for patients with liver metastasis; Renal function: serum creatinine ≤ 1.5 × ULN, or creatinine clearance (Ccr) ≥ 50 mL/min (Calculated according to the Cockcroft-Gault formula); Cockcroft-Gault formula: female Ccr (mL/min) = 0.85 × weight (kg) × (140-age)/ [72 × creatinine (mg/dL)] Coagulation function: international normalized ratio (INR) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

  13) Women of childbearing age are willing to take effective contraception from signing the ICF to 6 months after the last administration of the investigational drug. Women of childbearing age must have a negative blood pregnancy test result 7 days before the first dose.

Exclusion Criteria:

* 1) Pregnant or lactating women. 2) Active inflammatory breast cancer. 3) Previous treatment with other PARP inhibitor drugs, including but not limited to TSL-1502, Olaparib, Talazoparil, Fluzoparil, Nilaparib, Rucaparib, Veliparib, etc. 4) Known to be allergic to TSL-1502 or any excipient of TSL-1502 capsules. 5) Known to have active brain metastases (defined as meeting any of the following: stable neurological imaging < 4 weeks; symptoms related to brain metastasis; steroid therapy required; leptomeningeal disease); patients must have completed any prior treatment for brain metastases ≥ 4 weeks prior to the first dose.

  6) Patients with previous or current another malignancy. 7) Have other serious or uncontrollable clinical diseases or past medical history, surgical history, including but not limited to hepatic/renal dysfunction, respiratory disorders, endocrine disorders, metabolic disorders, neuropathy, or mental disorders, organ transplantation, etc.

  8) Gastrointestinal or digestive system diseases that may affect the absorption of investigational products as judged by the investigator or past medical history, such as intractable hiccups, nausea, vomiting, chronic gastrointestinal disease (e.g. Ron's disease, ulcerative colitis, active gastric ulcer, etc.), dysphagia, etc.

  9) Have serious cardiovascular system disease or past medical history (meet any of the following conditions); Definite cardiovascular abnormality within 6 months prior to first dose (e.g., myocardial infarction, cardiac arrhythmia, angina pectoris, angioplasty, vascular stent implantation, coronary artery bypass surgery, congestive heart failure, etc.); Baseline electrocardiogram QT or Fridericia-corrected QT interval (QTcF) prolongation [QTcF = QT/(RR 0.33), QTcF > 480 ms]; Left ventricular ejection fraction < 50% by cardiac ultrasound; Uncontrolled hypertension (Patients with blood pressure ≥150/100 mmHg after lifestyle improvement and medication) 10) Participated in clinical trials of other drugs or medical devices within 4 weeks prior to initial administration (note: except for those who did not use investigational drugs or medical devices).

  11) Patients who underwent major surgery or significant traumatic injury within 4 weeks prior to initial administration, or who planned to undergo major surgery in the trial period.

  12) Chemotherapy, radiotherapy, non-hormone targeted therapy, endocrine therapy, Anti-neoplastic immunotherapy [physiologic replacement doses of corticosteroids permitted (prednisone or equivalent < 15 mg/day)], Chinese medicine therapy with a clear indication for the treatment of breast cancer, or other anti-tumor therapy were received within 4 weeks prior to initial administration.

  13) AEs related to previous surgery and previous anti-tumor therapy (CTCAE version 5.0) did not recover to ≤ 1 grade (alopecia, pigmentation, platinum-induced neurotoxicity grade 2 and lower, except for clinically significant or asymptomatic laboratory abnormalities).

  14) Patients who had received a CYP2D6 liver enzyme inhibitors or inducers within 2 weeks prior to initial dosing, or who cannot discontinue the use of CYP2D6 liver enzyme inhibitors or inducers during the trial.

  15) Patients who test positive for treponema pallidum antibody, human immunodeficiency virus (HIV) antibody, hepatitis C virus (HCV) RNA, or active hepatitis B patients [defined as hepatitis B virus (HBV) DNA ≥ ULN].

  16) The investigator considered that patients have other conditions that might affect compliance or are not suitable for participating in this trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Radiological scans performed at baseline then every 6 weeks thereafter until objective radiological disease progression. Assessed up to a maximum of 40 months
  Defined as the proportion of patients with complete response (CR) and partial response (PR). Solid tumors evaluation criteria (RECIST) version 1.1 is used for anti-tumor efficacy evaluation. For patients with PR or CR at the first evaluation, response confirmation should be performed at least 4 weeks later

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | Radiological scans performed at baseline then every 6 weeks there after until disease progression or death due to any cause.Assessed up to a maximum of 40 months
  DCR is defined as the proportion of patients with CR, PR and stable disease (SD).
Duration of Response(DOR) | Radiological scans performed at baseline then every 6 weeks there after until disease progression or death due to any cause.Assessed up to a maximum of 40 months
  DOR is defined as the time from the first assessment of CR or PR to disease progression or death due to any cause.
Progress Free Survival(PFS) | Radiological scans performed at baseline then every 6 weeks there after until disease progression or death due to any cause.Assessed up to a maximum of 40 months
  PFS is defined as the time from randomization to the first disease progression or death due to any cause, whichever occurs first. 12 Months PFS Rate is defined as the percentage of subjects without disease progression or death from any cause 12 months after the beginning of randomization or the probability estimated by Kaplan-Meier method.
Overall Survival(OS) | Radiological scans performed at baseline then every 6 weeks there after until disease progression or death due to any cause.Assessed up to a maximum of 40 months
  OS is defined as the time from randomization to death due to any cause.
12 Months PFS Rate | Radiological scans performed at baseline then every 6 weeks there after until disease progression or death due to any cause.Assessed up to a maximum of 40 months
  12 Months PFS Rate is defined as the percentage of subjects without disease progression or death from any cause 12 months after the beginning of randomization or the probability estimated by Kaplan-Meier method.
Safety endpoints | From screening until final visit.Assessed up to a maximum of 40 months
  all AEs and SAEs by CTCAE v5.0

OTHER OUTCOMES:
Cmax | Cycle1(Day1、Day8、Day14 and Day21)
  Plasma concentrations for TSL-1502 and TSL-1502M will be analyzed to determine the maximum observed concentration
Cmin | Cycle1(Day1、Day8、Day14 and Day21)
  Plasma concentrations for TSL-1502 and TSL-1502M will be analyzed to determine the minimum observed concentration
AUC0-t | Cycle1(Day1、Day8、Day14 and Day21)
  Plasma concentrations for TSL-1502 and TSL-1502M will be analyzed to determine the area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Study Director — Jiangsu Tasly Diyi Pharmaceutical Co., Ltd.
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No